CLINICAL TRIAL: NCT00627458
Title: Immunogenicity and Reactogenicity of GSK Biologicals' DTPa-HBV-IPV/Hib Vaccine When Given as a Booster Dose
Brief Title: Immunogenicity and Reactogenicity of a Booster Dose of GSK Bio's DTPa-HBV-IPV/Hib Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111344
Record Dates: First submitted 2008-02-20; First posted 2008-03-03 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Acellular Pertussis; Diphtheria; Poliomyelitis; Haemophilus Influenzae Type b; Tetanus; Hepatitis B
Keywords: Hexavalent vaccine; Booster
MeSH Terms: conditions — Diphtheria; Poliomyelitis; Haemophilus Infections; Tetanus; Hepatitis B | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (3):
- INFANRIX HEXA PF GROUP (Experimental): Healthy male and female subjects between, and including 16 and 20 months of age at the time of booster vaccination, who were given the preservative-free (PF) formulation of Infanrix Hexa™ in the primary vaccination study 106786, additionally received a single booster dose of Infanrix Hexa™ vaccine, administered intramuscularly into the anterolateral quadrant of the right thigh.
  Interventions: Biological: Infanrix Hexa
- INFANRIX HEXA PC GROUP (Experimental): Healthy male and female subjects between, and including 16 and 20 months of age at the time of booster vaccination, who were given the preservative-containing (PC) formulation of Infanrix Hexa™ in the primary vaccination study 106786, additionally received a single booster dose of Infanrix Hexa™ vaccine, administered intramuscularly into the anterolateral quadrant of the right thigh.
  Interventions: Biological: Infanrix Hexa
- CONTROL GROUP (Active Comparator): Healthy male and female subjects between, and including 16 and 20 months of age at the time of booster vaccination, who were given the licensed formulation of Infanrix Hexa™ in the primary vaccination study 106786, additionally received a single booster dose of Infanrix Hexa™ vaccine, administered intramuscularly into the anterolateral quadrant of the right thigh.
  Interventions: Biological: Infanrix Hexa

INTERVENTIONS:
Biological: Infanrix Hexa — Vaccine administered as a booster dose at 16-20 months of age
  Other Names: GSK Biological's combined DTPa-HBV-IPV/Hib vaccine

SUMMARY:
The purpose of this booster study is to evaluate, in subjects primed in the primary study 106786, the persistence, at the time of the booster vaccination, of antibodies elicited by the different formulation of DTPa-HBV-IPV/ Hib vaccine (Infanrix Hexa TM). The study will also evaluate the immune response of these subjects to a DTPa-HBV-IPV/Hib booster. This protocol posting deals with the objectives and outcome measures of the booster phase. The objectives and outcomes measures of the primary phase are presented in a separate protocol posting (NCT = 00376779).

DETAILED DESCRIPTION:
This protocol posting has been updated in order to comply with the FDA AA, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol
* Subjects must have completed the full three-dose primary vaccination course with one of the formulations of the DTPa-HBV-IPV/Hib vaccine in primary study 106786.
* A male or female between, and including, 16 and 20 months of age at the time of booster vaccination.
* Written informed consent obtained from the parent or guardian of the subject
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose.
* Participation in another clinical study, between the primary study 106786 and the present booster study, or at any time during the study, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Planned administration or administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the administration of the booster dose and ending 30 days after the booster dose.
* Evidence of previous diphtheria, tetanus, pertussis, polio, hepatitis B and/or Hib booster vaccination or disease since the conclusion visit of study 106786.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.

Ages: 16 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 403 (Actual)
Dates: Start 2008-02-01; Primary Completion 2008-08-18 (Actual); Study Completion 2008-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Finland (6):
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111344 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix Hexa PF Group: Healthy male and female subjects between, and including 16 and 20 months of age at the time of booster vaccination, who were given the preservative-free (PF) formulation of Infanrix Hexa in the primary vaccination study 106786, additionally received a single booster dose of Infanrix Hexa vaccine, administered intramuscularly into the anterolateral quadrant of the right thigh.
- Infanrix Hexa PC Group: Healthy male and female subjects between, and including 16 and 20 months of age at the time of booster vaccination, who were given the preservative-containing (PC) formulation of Infanrix Hexa in the primary vaccination study 106786, additionally received a single booster dose of Infanrix Hexa vaccine, administered intramuscularly into the anterolateral quadrant of the right thigh.
- Control Group: Healthy male and female subjects between, and including 16 and 20 months of age at the time of booster vaccination, who were given the licensed formulation of Infanrix Hexa in the primary vaccination study 106786, additionally received a single booster dose of Infanrix Hexa vaccine, administered intramuscularly into the anterolateral quadrant of the right thigh.
Period: Overall Study
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
Started | 127 | 137 | 139
Completed | 123 | 130 | 133
Not Completed | 4 | 7 | 6
Not completed — Migrated from study area | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 6 | 5
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group | Total
Number analyzed (Participants) | 127 | 137 | 139 | 403
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.9 (1.12) | 18 (1.03) | 17.8 (1.11) | 17.90 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 66 | 59 | 181
  Male | 71 | 71 | 80 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: White-Caucasian/European heritage | 125 | 134 | 135 | 394
  Geographic ancestry: White-Arabic/North African heritage | 0 | 1 | 1 | 2
  Geographic ancestry: Not specified | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Toxoids
Description: A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: Before the booster administration (At Month 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 117
Participants
  Anti-D | 22 | 35
  Anti-T | 93 | 103

2. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Toxoids
Description: A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations greater than or equal to (≥) 0.1 IU/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 113 | 119
Participants
  Anti-D | 112 | 118
  Anti-T | 113 | 118

3. Primary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface Antigen (HBs)
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 milli international units per milliliter (mIU/mL). Also reported are the number of participants with anti-HBs antibody concentrations ≥ 100 mIU/mL.
Time Frame: Before the booster vaccination (At Month 0)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 117
Participants
  Anti-HBs ≥ 10 mIU/mL | 106 | 112
  Anti HBs ≥ 100 mIU/mL | 55 | 54

4. Primary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface Antigen (HBs)
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL. Also reported are the number of participants with anti-HBs antibody concentrations ≥ 100 mIU/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 118
Participants
  Anti-HBs ≥ 10 mIU/mL | 110 | 117
  Anti HBs ≥ 100 mIU/mL | 105 | 113

5. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Type 1, Type 2 and Type 3
Description: A seroprotected subject was defined as a subject with anti-Polio 1, 2 and 3 antibody titers ≥ the value of 8.
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 117
Participants
  Anti-polio 1: number analyzed (Participants) | 110 | 117
  Anti-polio 1 | 67 | 76
  Anti-polio 2 | 48 | 51
  Anti-polio 3 | 58 | 77

6. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus Type 1, Type 2 and Type 3
Description: A seroprotected subject was defined as a subject with anti-Polio 1, 2 and 3 antibody titers ≥ the value of 8.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 117
Participants
  Anti-polio 1: number analyzed (Participants) | 111 | 117
  Anti-polio 1 | 110 | 117
  Anti-polio 2 | 110 | 117
  Anti-polio 3 | 111 | 117

7. Primary Outcome: Number of Seroprotected Subjects Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN)
Description: A seroprotected subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 117
Participants
  Anti-PT: number analyzed (Participants) | 109 | 112
  Anti-PT | 80 | 81
  Anti-FHA: number analyzed (Participants) | 110 | 112
  Anti-FHA | 106 | 107
  Anti-PRN | 81 | 86

8. Primary Outcome: Number of Seroprotected Subjects Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN)
Description: A seroprotected subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 113 | 119
Participants
  Anti-PT: number analyzed (Participants) | 111 | 119
  Anti-PT | 111 | 118
  Anti-FHA: number analyzed (Participants) | 112 | 119
  Anti-FHA | 112 | 118
  Anti-PRN: number analyzed (Participants) | 113 | 118
  Anti-PRN | 113 | 117

9. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (PRP)
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentrations greater than or equal to (≥) 0.15 micrograms per milliliter (µg/mL). Also reported are the number of participants with anti-PRP antibody concentrations ≥ 1.0 µg/mL.
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 117
Participants
  Anti-PRP ≥ 0.15μg/mL | 71 | 87
  Anti-PRP ≥ 1.0μg/mL | 15 | 23

10. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (PRP)
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentrations ≥ 0.15 µg/mL. Also reported are the number of participants with anti-PRP antibody concentrations ≥ 1.0 µg/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 119
Participants
  Anti-PRP ≥ 0.15 µg/mL | 112 | 119
  Anti-PRP ≥ 1.0 µg/mL | 111 | 117

11. Primary Outcome: Number of Subjects With a Vaccine Response to PT, FHA and PR
Description: Vaccine response was defined as the appearance of antibodies in subjects who were initially seronegative (S-) [i.e. with concentrations lower than (<) the cut-off value] or at least doubling of pre-vaccination antibody concentrations in subjects who were initially seropositive (S+) [i.e. with concentrations greater than (>) the cut-off value).
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 116
Participants
  Anti-PT, S-: number analyzed (Participants) | 29 | 31
  Anti-PT, S- | 29 | 30
  Anti-PT, S+: number analyzed (Participants) | 78 | 81
  Anti-PT, S+ | 78 | 81
  Anti-PT, Total: number analyzed (Participants) | 107 | 112
  Anti-PT, Total | 107 | 111
  Anti-FHA, S-: number analyzed (Participants) | 4 | 5
  Anti-FHA, S- | 4 | 4
  Anti-FHA, S+: number analyzed (Participants) | 105 | 107
  Anti-FHA, S+ | 104 | 106
  Anti-FHA, Total: number analyzed (Participants) | 109 | 112
  Anti-FHA, Total | 108 | 110
  Anti-PRN, S-: number analyzed (Participants) | 31 | 31
  Anti-PRN, S- | 31 | 30
  Anti-PRN, S+: number analyzed (Participants) | 81 | 85
  Anti-PRN, S+ | 81 | 85
  Anti-PRN, Total | 112 | 115

12. Primary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 117
IU/mL
  Anti-D | 0.064 [0.058 to 0.071] | 0.069 [0.062 to 0.076]
  Anti-T | 0.216 [0.184 to 0.254] | 0.248 [0.213 to 0.289]

13. Primary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 113 | 119
IU/mL
  Anti-D | 2.237 [1.877 to 2.666] | 2.242 [1.868 to 2.689]
  Anti-T | 9.799 [8.39 to 11.444] | 9.136 [7.838 to 10.648]

14. Primary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 117
EL.U/mL
  Anti-PT: number analyzed (Participants) | 109 | 112
  Anti-PT | 7.8 [6.7 to 9.1] | 7 [6.1 to 8.1]
  Anti-FHA: number analyzed (Participants) | 110 | 112
  Anti-FHA | 21.7 [18.1 to 25.9] | 22.1 [18.5 to 26.2]
  Anti-PRN | 8.6 [7.1 to 10.3] | 8.7 [7.3 to 10.2]

15. Primary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 113 | 119
EL.U/mL
  Anti-PT: number analyzed (Participants) | 111 | 119
  Anti-PT | 150.9 [132.9 to 171.2] | 117.1 [101.5 to 135]
  Anti-FHA: number analyzed (Participants) | 112 | 119
  Anti-FHA | 609.6 [534.1 to 695.7] | 533.7 [463 to 615.1]
  Anti-PRN: number analyzed (Participants) | 113 | 118
  Anti-PRN | 308.5 [261.3 to 364.2] | 311.7 [260.3 to 373.2]

16. Primary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 117
mIU/mL | 84.3 [65.7 to 108.2] | 86.2 [67.8 to 109.6]

17. Primary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 118
mIU/mL | 3291.7 [2373.6 to 4565] | 3528.1 [2546.1 to 4888.9]

18. Primary Outcome: Anti-poliovirus Type 1, Type 2 and Type 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 111 | 117
Titers
  Anti-polio 1: number analyzed (Participants) | 110 | 117
  Anti-polio 1 | 12.9 [10.3 to 16.3] | 15.2 [12.3 to 18.9]
  Anti-polio 2 | 9.1 [7.3 to 11.3] | 8.7 [7.2 to 10.5]
  Anti-polio 3 | 9.5 [7.9 to 11.6] | 16 [12.6 to 20.4]

19. Primary Outcome: Anti-poliovirus Type 1, Type 2 and Type 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 117
Titers
  Anti-polio 1: number analyzed (Participants) | 111 | 117
  Anti-polio 1 | 726.3 [560.4 to 941.4] | 942.4 [734.1 to 1209.7]
  Anti-polio 2 | 712.8 [529.1 to 960.4] | 812.9 [632.8 to 1044.3]
  Anti-polio 3 | 780 [591 to 1029.3] | 1145.8 [891.6 to 1472.5]

20. Primary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in micrograms per milliliter (µg/mL).
Time Frame: Before the booster vaccination (At Month 0)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 119
µg/mL | 0.249 [0.199 to 0.31] | 0.314 [0.252 to 0.392]

21. Primary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in µg/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group
Number analyzed (Participants) | 112 | 119
µg/mL | 36.866 [28.61 to 47.504] | 35.318 [27.447 to 45.445]

22. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Toxoids
Description: A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.1 IU/mL .
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 119
Participants
  Anti-D, M0: number analyzed (Participants) | 111
  Anti-D, M0 | 40
  Anti-D, M1 | 119
  Anti-T, M0: number analyzed (Participants) | 111
  Anti-T, M0 | 95
  Anti-T, M1 | 119

23. Secondary Outcome: Number of Seroprotected Subjects Against Hepatitis B Surface Antigen (HBs)
Description: as for outcome 4
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 118
Participants
  Anti-HBs ≥ 10 mIU/mL, M0: number analyzed (Participants) | 110
  Anti-HBs ≥ 10 mIU/mL, M0 | 106
  Anti-HBs ≥ 10 mIU/mL, M1 | 118
  Anti HBs ≥ 100 mIU/mL, M0: number analyzed (Participants) | 110
  Anti HBs ≥ 100 mIU/mL, M0 | 67
  Anti HBs ≥ 100 mIU/mL, M1 | 114

24. Secondary Outcome: Number of Seroprotected Subjects Against Poliovirus Type 1, Type 2 and Type 3
Description: A seroprotected subject was defined as a subject with anti-polio 1, 2 and 3 antibody titers ≥ the value of 8.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 113
Participants
  Anti-polio 1, M0: number analyzed (Participants) | 109
  Anti-polio 1, M0 | 84
  Anti-polio 1, M1 | 112
  Anti-polio 2, M0: number analyzed (Participants) | 109
  Anti-polio 2, M0 | 56
  Anti-polio 2, M1 | 112
  Anti-polio 3, M0: number analyzed (Participants) | 109
  Anti-polio 3, M0 | 82
  Anti-polio 3, M1 | 113

25. Secondary Outcome: Number of Seroprotected Subjects Against PT, FHA and PRN
Description: A seroprotected subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL .
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 119
Participants
  Anti-PT, M0: number analyzed (Participants) | 110
  Anti-PT, M0 | 93
  Anti-PT, M1 | 119
  Anti-FHA, M0: number analyzed (Participants) | 109
  Anti-FHA, M0 | 109
  Anti-FHA, M1 | 119
  Anti-PRN, M0: number analyzed (Participants) | 111
  Anti-PRN, M0 | 99
  Anti-PRN, M1 | 119

26. Secondary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (PRP)
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentrations ≥ 0.15 μg/mL. Also reported are the number of participants with anti-PRP antibody concentrations ≥ 1.0 µg/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 119
Participants
  Anti-PRP ≥ 0.15 μg/mL, M0: number analyzed (Participants) | 111
  Anti-PRP ≥ 0.15 μg/mL, M0 | 92
  Anti-PRP ≥ 0.15 μg/mL, M1 | 119
  Anti-PRP ≥ 1.0 μg/mL, M0: number analyzed (Participants) | 111
  Anti-PRP ≥ 1.0 μg/mL, M0 | 32
  Anti-PRP ≥ 1.0 μg/mL, M1 | 118

27. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in IU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Control Group
Number analyzed (Participants) | 119
IU/mL
  Anti-D, M0: number analyzed (Participants) | 111
  Anti-D, M0 | 0.084 [0.073 to 0.097]
  Anti-D, M1 | 3.952 [3.365 to 4.642]
  Anti-T, M0: number analyzed (Participants) | 111
  Anti-T, M0 | 0.261 [0.219 to 0.31]
  Anti-T, M1 | 10.833 [9.505 to 12.347]

28. Secondary Outcome: Anti-PT, Anti-FHA, Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Control Group
Number analyzed (Participants) | 119
EL.U/mL
  Anti-PT, M0: number analyzed (Participants) | 110
  Anti-PT, M0 | 8.9 [7.7 to 10.3]
  Anti-PT, M1 | 153.7 [135.1 to 174.9]
  Anti-FHA, M0: number analyzed (Participants) | 109
  Anti-FHA, M0 | 33.7 [27.6 to 41.1]
  Anti-FHA, M1 | 791.9 [708.8 to 884.8]
  Anti-PRN, M0: number analyzed (Participants) | 111
  Anti-PRN, M0 | 15.3 [12.6 to 18.5]
  Anti-PRN, M1 | 564.1 [489.5 to 650.1]

29. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Control Group
Number analyzed (Participants) | 118
mIU/mL
  Anti-HBs, M0: number analyzed (Participants) | 110
  Anti-HBs, M0 | 139.8 [107.2 to 182.3]
  Anti-HBs, M1 | 6132.7 [4587.8 to 8197.9]

30. Secondary Outcome: Anti-poliovirus Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Control Group
Number analyzed (Participants) | 113
Titers
  Anti-polio 1, M0: number analyzed (Participants) | 109
  Anti-polio 1, M0 | 21.6 [17.1 to 27.4]
  Anti-polio 1, M1 | 1288.8 [1029.1 to 1614]
  Anti-polio 2, M0: number analyzed (Participants) | 109
  Anti-polio 2, M0 | 11.8 [9.2 to 15]
  Anti-polio 2, M1 | 1231 [961 to 1576.9]
  Anti-polio 3, M0: number analyzed (Participants) | 109
  Anti-polio 3, M0 | 21.3 [16.4 to 27.7]
  Anti-polio 3, M1 | 1794.8 [1426.8 to 2257.7]

31. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in µg/mL.
Time Frame: Before (Month 0) and one month after (Month 1) the booster vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Control Group
Number analyzed (Participants) | 119
µg/mL
  Anti-PRP, M0: number analyzed (Participants) | 111
  Anti-PRP, M0 | 0.487 [0.383 to 0.62]
  Anti-PRP, M1 | 77.087 [60.224 to 98.672]

32. Secondary Outcome: Number of Subjects With a Vaccine Response to PT, FHA and PR
Description: Vaccine response was defined as the appearance of antibodies in subjects who were initially seronegative (S-) (i.e. with concentrations < cut-off value) or at least doubling of pre-vaccination antibody concentrations in subjects who were initially seropositive (S+) (i.e. with concentrations > cut-off value).
Time Frame: One month after the booster dose (At Month 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group
Number analyzed (Participants) | 111
Participants
  Anti-PT, S-: number analyzed (Participants) | 17
  Anti-PT, S- | 17
  Anti-PT, S+: number analyzed (Participants) | 93
  Anti-PT, S+ | 93
  Anti-PT, Total: number analyzed (Participants) | 110
  Anti-PT, Total | 110
  Anti-FHA, S-: number analyzed (Participants) | 0
  Anti-FHA, S- | 0
  Anti-FHA, S+: number analyzed (Participants) | 109
  Anti-FHA, S+ | 105
  Anti-FHA, Total: number analyzed (Participants) | 109
  Anti-FHA, Total | 105
  Anti-PRN, S-: number analyzed (Participants) | 12
  Anti-PRN, S- | 12
  Anti-PRN, S+: number analyzed (Participants) | 99
  Anti-PRN, S+ | 98
  Anti-PRN, Total | 110

33. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after the booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with their symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
Number analyzed (Participants) | 126 | 136 | 138
Participants
  Any Pain | 74 | 76 | 82
  Any Redness | 66 | 79 | 94
  Any Swelling | 44 | 53 | 60

34. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as rectal temperature equal to or above (≥) 38.0 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after the booster vaccination
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
Number analyzed (Participants) | 126 | 136 | 138
Participants
  Any Drowsiness | 50 | 48 | 58
  Any Fever (Rectal) | 22 | 34 | 31
  Any Irritability | 68 | 86 | 78
  Any Loss of Appetite | 37 | 46 | 45

35. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-30) follow-up period after the booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
Number analyzed (Participants) | 127 | 137 | 139
Participants | 51 | 54 | 61

36. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Assessed SAEs include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 1, during the entire study period
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
Number analyzed (Participants) | 127 | 137 | 139
Participants | 1 | 2 | 1

37. Secondary Outcome: Number of Subjects Reporting Concomitant Medications
Time Frame: During the 4-day (Days 0-3) follow-up period after the booster vaccination
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
Number analyzed (Participants) | 127 | 137 | 139
Participants
  Any concomitant medication | 105 | 111 | 116
  Any antipyretic | 34 | 35 | 33

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) period after the booster vaccination. Unsolicited AEs: during the 31-day (Days 0-30) period after the booster vaccination. SAEs: during the entire study period (from Month 0 up to Month 1).
Arm/Group | Infanrix Hexa PF Group | Infanrix Hexa PC Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/137 | 0/139
Serious Adverse Events (participants affected / at risk) | 1/127 | 2/137 | 1/139
Other Adverse Events (participants affected / at risk) | 116/127 | 126/137 | 129/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix Hexa PF Group (N=127) | Infanrix Hexa PC Group (N=137) | Control Group (N=139)
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia adenoviral (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infanrix Hexa PF Group (N=127) | Infanrix Hexa PC Group (N=137) | Control Group (N=139)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 0
Pain (General disorders) | 74/126 | 76/136 | 82/138
Redness (General disorders) | 66/126 | 79/136 | 94/138
Swelling (General disorders) | 44/126 | 53/136 | 60/138
Drowsiness (General disorders) | 50/126 | 48/136 | 58/138
Fever/(Rectal) (General disorders) | 22/126 | 34/136 | 31/138
Irritability (General disorders) | 68/126 | 86/136 | 78/138
Loss of appetite (General disorders) | 37/126 | 46/136 | 45/138
Pyrexia (General disorders) | 6 | 5 | 8
Injection site induration (General disorders) | 5 | 2 | 10
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 5
Otitis media (Infections and infestations) | 4 | 7 | 14
Upper respiratory tract infection (Infections and infestations) | 9 | 8 | 6
Rhinitis (Infections and infestations) | 3 | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.